CLINICAL TRIAL: NCT05765214
Title: Impact of Colorectal Cancer and Nutrition Education Program Among Minority Patients With Type 2 Diabetes
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charles Drew University of Medicine and Science (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: G003CSG1
Record Dates: First submitted 2023-03-01; First posted 2023-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer; Type 2 Diabetes
Keywords: nutrition education
MeSH Terms: conditions — Colorectal Neoplasms; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (IG) (Experimental): Participants randomized to the IG will receive a customized patient-centered, culturally appropriate education program. Patients randomized to the IG will participate in eight (8) education sessions. A booklet with colorectal cancer education and nutrition education will be developed and print materials given to the participants to use as a workbook.
  Interventions: Behavioral: Intervention Group (IG)
- Usual Care (UC) (No Intervention): Patients randomized to UC group will continue to receive care at the clinic without any intervention from the study team.

INTERVENTIONS:
Behavioral: Intervention Group (IG) — In general, the education will cover:
  (i) Colorectal cancer - knowledge, perceptions, self-care, and social norms (CRC-KPSS): Knowledge; Perceptions (perceived susceptibility, perceived severity, perceived benefits, perceived barriers); Self-care; and Social norms; and information on colorectal cancer screening (ii) Healthy nutrition colorectal for cancer risk reduction and complementary to diabetes guideline (increasing consumption of fiber, fruits, vegetables, whole grains, and calcium; reducing red and processed meat, fat, added sugars and alcohol)
  Arms: Intervention Group (IG)

SUMMARY:
The goal of this observation study is to deliver an education program designed to increase knowledge of colorectal cancer prevention and nutrition education in minorities with Type 2 diabetes. The main questions it aims to answer are:

* What factors are associated with colorectal cancer screening among patients with type 2 diabetes?
* Will implementing a customized patient-centered, culturally appropriate colorectal cancer education, and nutrition education program reduce the risk for colorectal cancer among patients with type 2 diabetes?
* What is the impact of a patient-centered, culturally appropriate colorectal cancer education, and nutrition education intervention program on colorectal cancer screening and dietary indices among patients with type 2 diabetes compared to outcomes with patients who do not receive the intervention (usual care)?

Participants randomized to the intervention group will:

* receive a customized patient-centered, culturally appropriate education program
* participate in eight (8) education sessions
* be given booklet with colorectal cancer education and nutrition education to use as a workbook

Researchers will compare colorectal cancer knowledge, perceptions, self-care, and social norms scores and dietary indices of the intervention group to the control group immediately and 6-months post intervention to see if the education program increased colorectal cancer knowledge and screenings and changes in dietary habits.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the second leading cause of death in the United States (US)1. In 2019, over 140,000 adults were newly diagnosed with CRC and over 50,000 died.Furthermore, colorectal cancer disproportionately affects minorities and individuals with diabetes. Research has proven that interventions can increase cancer screening rates and improve lifestyle choices that put minorities at higher risk for developing colorectal cancer and diabetes.

This proposal will assess the impact of a colorectal cancer and nutrition education program among minority patients with type 2 diabetes by carrying out three aims.

Aim 1: Examine factors associated with colorectal cancer screening among patients with type 2 diabetes. The aim of this objective is to identify factors associated with colorectal cancer screening among patients with type 2 diabetes by comparing patients who have received screening verses those who have not. It is hypothesized that patients with type 2 diabetes who have not met colorectal cancer screening guidelines have low socioeconomic status (income 100% below poverty level, lack health insurance, speak language other than English, less education); have fewer provider visits; are not married; and have poor health and health risk factors (uncontrolled diabetes, multiple comorbidities (3+), BMI>30, depression, smoking and alcohol use history) compared to patients with type 2 diabetes who have met screening guidelines.

Aim 2:Implement a customized patient-centered, culturally appropriate colorectal cancer education, and nutrition education program aimed at reducing the risk for colorectal cancer among patients with type 2 diabetes at a community health center. The aim of this objective is to deliver a customized patient-centered, culturally appropriate education program on (i) colorectal cancer (knowledge, perceptions, self-care, social norms; and colorectal cancer screening) and (ii) healthy nutrition based on dietary guidelines for colorectal cancer risk reduction and complementary to type 2 diabetes dietary guidelines, among minority patients at a community health center.

Aim 3: Assess the impact of a patient-centered, culturally appropriate colorectal cancer education, and nutrition education intervention program on colorectal cancer screening and dietary indices among patients with type 2 diabetes; and compare outcomes with patients who do not receive the intervention (usual care). The first objective of this aim is to measure change in knowledge and perceptions about colorectal cancer, and colorectal cancer screening immediately and 6 months post intervention. It is hypothesized that patients in the intervention group will have (1) higher knowledge and higher perception scores compared to those receiving usual care and (2) 25% higher rate of colorectal cancer screening 12 months after the intervention, compared to those receiving usual care. The aim's second objective is to measure the change in dietary indices associated with colorectal cancer (fiber, fruits, vegetables, calcium, red meat, processed meat, fat, and alcohol consumption)and overall diet quality immediately and 6 months post intervention. It is hypothesized that patients who receive a patient-centered culturally appropriate nutrition education intervention program will be more likely to meet dietary guidelines for fiber, fruits, vegetables, calcium, red meat, processed meat, fat, and alcohol consumption and overall diet quality compared those receiving usual care.

A five-phase study will be carried out at the Kedren Community Health Center (KCHC) in South Los Angeles that had a patient population of 48.4% African American and 47.5% Hispanic in 2020. Surveys and electronic health record will be used to recruit patients and provide study data. The impact of an education program will be assessed by comparing an intervention verses a control group, and change in knowledge, perceptions, and behaviors related to nutrition and colorectal cancer screening over time.

A major anticipated outcome is increasing the rate of colorectal cancer screening among diabetic patients at KCHC. Another outcome is improving dietary choices among study participants. One or more manuscripts will be prepared for publication and findings will be presented at professional conferences and community forums.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes type 2 diagnosis
* Age 35-75
* Any gender
* African American race (Hispanic or non-Hispanic)
* Hispanic ethnicity (any race)
* Have had at least one visit to KCHC in the past 2 years
* Have complete address and telephone number in the electronic health records. Although USPSTF and American Cancer Society screening guidelines recommend starting screening at age 45, our intervention will include patients age 35-44 due to the reported incidence of CRC at an earlier age among diabetic patients 3

Exclusion Criteria:

* History of colorectal cancer
* History of colectomy
* History of colonic polyps (ICD-10 Z86.010)
* History of radiation treatment for another cancer (abdominal prostate, skin etc)
* History of Crohn's disease
* Ulcerative colitis
* Cystic fibrosis
* <10 year life expectancy
* Cognitive impairment or inability to comprehend or provide consent to participate in the study
* Being institutionalized
* Participating in another diet program

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
CRC-KPSS change and screening uptake | immediately and 6-months post-intervention
  Change in colorectal cancer knowledge, perceptions, self-care, and social norms; improved dietary quality and change in colorectal cancer screening uptake

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Kibe, DrPH, Principal Investigator — Charles Drew University of Medicine and Science
Locations (1):
- Charles R. Drew University, Los Angeles, California, United States